CLINICAL TRIAL: NCT04180917
Title: Current Trends and Future Perspectives Regarding Elective Rotations Abroad Within Italian Surgical Residency Training: Is the Glass Half Empty or Half Full?
Brief Title: Current Trends and Future Perspectives Regarding Elective Rotations
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianluca Costa, Clinical Professor, MD, PhD, University of Roma La Sapienza
Other Study IDs: Ita-SURG_S_2019
Record Dates: First submitted 2019-10-30; First posted 2019-11-29 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Surgery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — survey

SUMMARY:
Surgical resident elective rotation abroad give different opportunity such experience a different teaching and training, acquire more and new operative experience, experience living and working in a different cultural environment. Furthermore, the growing process of globalization that involves the nations themselves in different sectors, should also lead to a homogeneity of training on a global level, in order to be able to guarantee adequate assistance to different types of patients at the same time, and the possibility for doctors themselves of working abroad. the objective of the study is to provide the first overview of what is the current Italian scenario concerning abroad elective rotations during surgical training

ELIGIBILITY:
Inclusion Criteria:

* working as short-term supernumerary registrars in a foreign surgical department during the academic year 2017-2018

Exclusion Criteria:

* Surgeons/residents who have not been abroad for training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: resident
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction grade of actual elective rotation abroad in Italy | 1 years
  A five point Likert-type scale

SECONDARY OUTCOMES:
Gender | 1 year
  Ratio male/gender
Age at time of elective training | 1 year
  Age
Year of residency at the time of elective training | 1 year
  Multiple choice answers accounting 1 to 6
Institution visited | 1 year
  Multiple choice accounting 5 option such as university hospital, tertiary care hospital, referral center
Global surgical exposure | 1 year
  A five point Likert-type scale

IPD SHARING:
Plan to Share IPD: No
no one